CLINICAL TRIAL: NCT02566538
Title: Prospective Population Based Cohort Study on Cognitive and Cardiovascular Aging
Brief Title: Prospective Population Based Cohort Study on Cognitive and Cardiovascular Aging (MonaLisaPredor)
Acronym: MLP
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC31/12/0400; 2012-A00943-40 (Other: ANSM, ID-RCB)
Record Dates: First submitted 2013-05-24; First posted 2015-10-02 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Aging
Keywords: Cohort study; psychometric tests; cognitive function; cardiovascular risk; prediction algorithm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Aging is a long term process, starting early in life, and progressively affecting various functions and organs. Cardiovascular diseases and cognitive impairment are two conditions related to advancing age and sharing common risk factors. The Mona Lisa- PREDOR study is a population-based prospective cohort study carried out to develop risk prediction algorithms aimed at identifying people who are the most likely to develop impaired psychometric and cognitive functioning and impaired cardiovascular risk, in the coming years.

DETAILED DESCRIPTION:
The study is aimed at identifying predictors of impaired changes in psychometric and cognitive performances and level of cardiovascular risk, over a seven-year period, and to develop risk prediction algorithms. Main secondary objectives are to study response to psychometric and cognitive tests according to age, and to estimate the prevalence of the frailty syndrome according to age.

The design is a prospective cohort study carried out among 1500 men and women from the general population, aged 42-89 years, and living in South-western France. Except for participants aged 80-89 years, all participants have been previously assessed in 2005-2007, as regard to their psychometric and cognitive performances and level of cardiovascular risk, as part of the Mona Lisa study.

Data collection includes a detailed questionnaire on previous medical history, drug intake, education level, and life habits; a standardised clinical examination; psychometric tests (word list learning test, digit symbol substitution test, word fluency test and Stroop test), and a fasting blood sample. Level of cardiovascular risk and frailty syndrome were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 42-79 years, living in South-western France, who participated in the Mona Lisa Study (2005-2007) (in the Mona Lisa study, participants were selected by drawing on polling lists)
* Men and women aged 80-89 years, living in South-western France, selected by drawing on polling lists.

Exclusion Criteria:

* Subject who refuses to participate (who refuses to sign the inform consent)
* Subject not affiliated to a health assurance system
* Subject with altered cognitive functioning compromising the understanding of the information on the study, and not accompanied by a trusted third party.

Ages: 42 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The design is a prospective cohort study carried out among 1500 men and women from the general population, aged 42-89 years,and living in South-western France. Except for participants aged 80-89 years, all participants have been previously assessed in 2005-2007, as regard to their psychometric and cognitive performances and level of cardiovascular risk, as part of the Mona Lisa study.
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2013-05-22 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Test of memorizing and restitution of words | 7 years after the first assessment
  French version of the Rey auditory verbal learning test

SECONDARY OUTCOMES:
Level of cardiovascular risk | 7 years after the first assessment
  Number of risk factors
Level of cardiovascular risk | 10 years after the first assessment
  10-years risk of cardiovascular event. A first assessment was performed in 2005-2007. A second one will be performed as part of the current study (2013-2016).
WAIS-DSST | 7 years after the first assessment
  Wechsler Adult Intelligence Survey - Digit Symbol Substitution Subtest
Stroop test | 7 years after the first assessment

CONTACTS AND LOCATIONS:
Overall Officials: Vanina BONGARD, MD, PhD, Principal Investigator — University Hospital, Toulouse; Jean FERRIERES, MD PhD, Study Chair — University Hospital, Toulouse; Bruno VELLAS, MD PhD, Study Chair — University Hospital, Toulouse; Jean-Bernard RUIDAVETS, MD, Study Chair — University Hospital, Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, France